CLINICAL TRIAL: NCT04302597
Title: Cosmetic Outcomes After Skin Closure of Pfannenstiel Incision With Tissue Adhesive (2-octylcyanoacrylate) or Staples in Repeated Cesarean Section
Brief Title: Cosmetic Outcomes With Tissue Adhesive (2-octylcyanoacrylate) or Staples in Repeated Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLUE-1
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Section
Keywords: Cesarean delivery; Cosmesis; Healing; Skin closure; Scar assessment scales
MeSH Terms: interventions — Sutures; Tissue Adhesives

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staples (Active Comparator): Women who underwent repeated cesarean section with skin closure using staples.
  Interventions: Procedure: Staples
- Tissue adhesive (Experimental): Women who underwent repeated cesarean section with skin closure using 2-octylcyanoacrylate tissue adhesive.
  Interventions: Procedure: Tissue adhesive

INTERVENTIONS:
Procedure: Staples — Skin closure using surgical stapler.
  Arms: Staples
Procedure: Tissue adhesive — Skin closure using 2-octylcyanoacrylate tissue adhesive.
  Arms: Tissue adhesive

SUMMARY:
Recent clinical trials were developed to test the outcomes of skin closure with tissue adhesive, staples and monofilament synthetic suture after cesarean section with Pfannenstiel incision: both clinical outcomes such as blood loss, surgical site infection, length of postpartum hospitalization, or wound disruption, as well as Patient and Observer Scar Assessment Scale (POSAS) scores 8 weeks after surgery, were comparable between these different skin closure methods.

Despite the available studies are often based on robust methodologies and appropriate assessment scales, most of them were aimed to evaluate cosmetic outcomes in primary cesarean section, whereas data analyses published so far do not allow to draw a firm conclusion about repeated cesarean sections. Based on these elements, the aim of this study is to evaluate cosmetic outcomes after skin closure of Pfannenstiel incision with tissue adhesive or staples in a selected population undergoing repeated cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Previous cesarean section with Pfannenstiel incision (regardless of the indication, emergency/urgency, weeks of pregnancy and years passed from the previous cesarean section)
* Maternal age 18-45 years
* Singleton pregnancy at 37-41 weeks of gestation (based on first-trimester ultrasound) with a viable fetus

Exclusion Criteria:

* History of keloids
* Previous transversal suprapubic scars
* Clinical signs of infection and/or tattoos in the area to be studied
* Known patient hypersensitivity to any of the suture materials used in the protocol
* BMI below 20 or above 30
* Any medical disorder that could affect wound healing, including severe malnutrition, conditions requiring chronic corticosteroid use or immune suppressant, uncontrolled diabetes mellitus (defined as Hemoglobin A1c > 6%, unbalanced daily glucose measurements, and fasting glucose >95 mg/dL).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Observer Scar Assessment Scale (OSAS) score | 6 months after repeated cesarean section
  The Observer Scar Assessment Scale (OSAS) rates 5 variables: vascularity, pigmentation, thickness, relief, and pliability. Each variable uses a 10-point scoring system, with 1 representing normal skin. Ratings of individual variables may be summed to obtain a total score ranging from 5-50, with 5 representing normal skin.

SECONDARY OUTCOMES:
Patient Scar Assessment Scale (PSAS) score | 6 months after repeated cesarean section
  The Patient Scar Assessment Scale (PSAS) consists of 6 items on scar-related pain, itchiness, color, stiffness, thickness, and irregularity. Each item uses a 10-point scoring system, summed to obtain a total score ranging from 6-60, with 6 representing normal skin with no associated symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Cromi, M.D., Ph.D., Principal Investigator — Università degli Studi dell'Insubria; Fabio Ghezzi, M.D., Study Chair — Università degli Studi dell'Insubria; Antonio Simone Laganà, M.D., Ph.D., Study Chair — Università degli Studi dell'Insubria
Locations (1):
- Ospedale "Filippo Del Ponte", Varese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No